CLINICAL TRIAL: NCT05054491
Title: Evaluation of the Feasibility, Acceptability and Impact of Group-based Antenatal Care at the Health Post Level on Continuation in Antenatal Care and Facility-based Delivery in Amhara, Ethiopia Using a Cluster Randomized Step-wedge Design
Brief Title: Ethiopia Group Antenatal Care Study at the Health Post Level
Acronym: ARC004
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We are not able to continue the study as there is conflict in the study area that prevents women from gathering for group antenatal care. It is also not safe for data collectors to collect data in the study sites.
Sponsor: Jhpiego (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Addis Continental Institute of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 14448
Record Dates: First submitted 2021-08-11; First posted 2021-09-23 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Antenatal Care
Keywords: Ethiopia; Health post; Group ANC

STUDY DESIGN:
Intervention Model Description: Stepped wedge design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ANC (Experimental): Intervention period in stepped wedge design where women are receiving antenatal care in a group setting
  Interventions: Behavioral: Group Antenatal Care
- Individual ANC (routine) (No Intervention): Pre-intervention time period (control period) where the intervention is not being implemented yet (women are receiving individual antenatal care as is currently offered)

INTERVENTIONS:
Behavioral: Group Antenatal Care — Group ANC is an integrated approach that incorporates physical assessment, education and skill development, and peer support and takes a broader, more holistic, woman-centered approach to traditional antenatal care
  Arms: Group ANC

SUMMARY:
The purpose of this study is to determine the acceptability, feasibility, and effectiveness of a group antenatal care (G-ANC) model introduced at the health post level compared to usual antenatal care (ANC) among women who report intention to receive ANC at the health post level.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 15 years at the time of enrollment; pregnant 15-17 year-olds will be treated as emancipated/mature as per local regulations
* Gestational age less than or equal to 20 weeks at the time of enrollment determined by last menstrual period (LMP), pelvic exam, fundal height, quickening, ultrasound, and/or timing of fetal heart tones and pregnancy test
* Pregnant women able and willing to provide adequate locator information
* Planning to reside at their current location for at least 10 months
* Agree to participate in the study and continue ANC at health post
* Willing to participate and consent to follow up for up to 6 weeks post-delivery
* Are willing to receive group antenatal care at the health post level (during the intervention period)

Exclusion Criteria:

* Women who plan to travel away from the study site for more than four consecutive weeks during ANC or after 6 weeks post-delivery
* Women who are unable provide consent
* Women who have any condition that in the opinion of the investigator or designee, would complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 540 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Acceptability of G-ANC at the health post level | Less than or equal to 20 weeks gestation at enrollment into study up to 6 weeks after delivery
  Satisfaction survey to understand satisfaction with G-ANC
Feasibility of G-ANC at the health post level | Less than or equal to 20 weeks gestation at enrollment into study up to 6 weeks after delivery
  Documentation of number of G-ANC sessions facilitated by by health extension workers to measure feasibility
Effectiveness of G-ANC on continuation of ANC | Less than or equal to 20 weeks gestation at enrollment into study up to 6 weeks after delivery
  Survey of self-reported number of ANC visits to document effectiveness of continuing ANC

SECONDARY OUTCOMES:
Effectiveness of G-ANC on quality of care | Less than or equal to 20 weeks gestation at enrollment into study up to 6 weeks after delivery
  Survey of self-reported quality of care elements received during ANC to understand role of G-ANC on improving elements of quality of care during ANC

CONTACTS AND LOCATIONS:
Locations (1):
- Enashenifalen, Mecha, North Mecha Woreda, West Gojam Zone, Amhara Region, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with the Gates ARC partner, RTI

REFERENCES:
- [Derived] Yallew WW, Fasil R, Berhanu D, Wolde K, Teshite D, Sethi R, Yenokyan G, Woldemariam Y, Suhowatsky S, Hyre A, Noguchi L, Worku A. Evaluation of the feasibility, acceptability, and impact of Group Antenatal Care at the health post level on continuation in antenatal care and facility based delivery in Ethiopia using a cluster randomized stepped-wedge design: Study protocol. Gates Open Res. 2025 Jan 31;8:29. doi: 10.12688/gatesopenres.15190.3. eCollection 2024. PMID 39936142